CLINICAL TRIAL: NCT01546766
Title: Developing a Non-invasive Method and Device for Assessing the Degree of Midperipheral Retinal Ischemia in Diabetic Retinopathy.
Brief Title: Rapid, Non-invasive, Regional Functional Imaging of the Retina. (Diabetic Retinopathy Diagnosis Device)
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Neurolign (Industry); Jules Stein Eye Institute (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Michael B. Gorin, Professor in Ophthalmology, University of California, Los Angeles
Other Study IDs: UCLA IRB#11-002987; 5R44EY018025-03 (NIH)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Diabetes; Retinal Disorders
Keywords: Diabetes; Pupillary response; Retinal disorders; Midperipheral ischemia; Fundus photography; Optical coherence tomography
MeSH Terms: conditions — Diabetes Mellitus; Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects with diabetes: (Subjects that have been diagnosed with diabetes).
  Interventions: Device: Pupillometry testing.
- Control volunteers: (Subjects with no history of ocular problems).
  Interventions: Device: Pupillometry testing.
- Subjects with retinal conditions: (Subjects with a history of retinal disorders except diabetes).
  Interventions: Device: Pupillometry testing.

INTERVENTIONS:
Device: Pupillometry testing.

SUMMARY:
The basic objective of this project is to test a modification of existing technology for monitoring the responses of the pupil to light as a method for detecting regional losses of function of the retina. The "instrument" consists of a commercially available set of goggles that monitor the eye positions and pupils using infrared light and small cameras. The signals from the monitoring cameras are collected in a computer that records how their pupils have responded to each lighting condition. Because diabetics develop damage initially to certain parts of the retina before they have more serious damage, the ultimate goal of this research is to develop a simple, noninvasive, rapid method for widespread screening of diabetics in order to identify those who may require medical attention and/or therapy for diabetic retinopathy.

DETAILED DESCRIPTION:
This study consists of three parts. The first part is to work with a limited number of normal individuals and those with known diabetic retinopathy to test a variety of the light conditions to find those that appear to be optimal for detecting retinal damage. The second part of this study, which is to test the instrument and these conditions with both normal subjects and a series of diabetics with varying degrees of severity of diabetic retinopathy. This part of the study is intended to determine how sensitive and specific the detection method is over the full range of retinal damage that is observed in diabetics. The third part of this study is to use the same instrument either with the same testing conditions as used for the diabetics or with modifications based on the regional areas of the retina that are damaged for other conditions, including (but not limited to) sickle cell retinopathy, retinitis pigmentosa, vascular diseases of the retina.

The risks from this study are minimal. All of the portions of the study that are required for the clinical assessment of the participant's retinal health are consistent with the standard of care for their condition. For diabetics with no clinically evident retinal damage from diabetes, they will receive a regular dilated eye exam and photographs to document the appearance of their retina. For those with more severe diabetic changes, special retinal photographs and fluorescein angiography (photographs taken in the presence of a dye that is injected into an arm vein that allows one to study the detailed changes of the blood vessels in the retina) will be done to more accurately assess the degree of diabetic damage.

The long-term objective of this application is to develop an imaging device for the early detection, diagnosis and quantification of the degree of midperipheral retinal ischemia in Diabetic Retinopathy (DR). Earlier diagnosis of DR could facilitate intervention at a stage that may prevent or lessen permanent damage from the ravages of the disease, in turn, improving patient quality of life and reducing lifetime treatment costs. DR is one of the more debilitating potential outcomes of diabetes posing a major threat to the quality of life of diabetics. Experts believe that DR is the leading cause of blindness in the industrialized world in people between the ages of 25 and 74 years old.

The American Academy of Ophthalmology states that DR is the leading cause of blindness among working Americans and currently affects nearly seven million people in the U.S. Early detection can help treat DR and salvage about 90 percent of vision loss, but about one-third of the diabetic population remains undiagnosed, translating into approximately 5.7 million people in the U.S. Delay in the primary diagnosis of diabetes allows diabetic complications to progress significantly before detection further increasing the risks associated with the disease by making the treatment much more complicated. Diabetes management guidelines advocate initiation of therapeutic intervention early in the prognosis of the disease. Estimates of diabetics in the U.S. with DR range from 15% to as high as 40%.

ELIGIBILITY:
Inclusion Criteria:

* All subjects: must be greater than 18 years of age and capable of understanding informed consent.
* All subjects must be willing to tolerate the placement of a set of goggles on their face.
* All subjects must have visual acuities of 20/60 or better in at least one eye.
* Normal subjects must have a history of a normal eye examination within one year prior to participation in this study.
* Normal subjects must have no history of ocular disease and no history of diabetes.
* Diabetic subjects must be diagnosed with diabetes upon prior clinical examination.
* Retinal Conditions subjects must be diagnosed with a retinal pathology, hereditary or acquired.

Exclusion Criteria:

* Subjects with glaucoma and high myopia are specifically excluded.
* Diabetic subjects may not have had laser (panretinal photocoagulation) in both eyes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 145 normal adults 270 adults with diabetic retinopathy 50 adults with retinal conditions
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2007-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pupillary response | 3 months
  We will analyze the following three components of the pupillary response: latency, constriction velocity and amplitude. The measurements will be taken after initiation of the light stimulus.
  These functions will be determined for each eye of each subject using both the central and annular stimuli. Each set of experimental conditions will yield a unique relative luminance ratio that can be used to compare the relative functional integrity of the peripheral retina with respect to the central macula.

SECONDARY OUTCOMES:
Pupillary response. | 1 year
  Constriction velocity, latency and amplitude will allow us to compare the sensitivity of the testing methods with a variety of diabetic cases so that we can establish the most appropriate method for generalized screening.
  The secondary measures will include the differences in maximal constriction and the pupil diameters at the time of maximal rate of constriction as well as analyses of the impact of the light stimuli on the three latency measures of response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Gorin, MD, PhD, Principal Investigator — Jules Stein Eye Institute, Dept. of Ophthalmology, David Geffen School of Medicine at UCLA; Alexander Kiderman, PhD, Study Director — Neuro Kinetics, Inc.
Locations (2):
- United States (2):
  - Jules Stein Eye Institute, Dept. of Ophthalmology, David Geffen School of Medicine at UCLA, Los Angeles, California
  - Neuro Kinetics Inc., Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Ortube MC, Kiderman A, Eydelman Y, Yu F, Aguilar N, Nusinowitz S, Gorin MB. Comparative regional pupillography as a noninvasive biosensor screening method for diabetic retinopathy. Invest Ophthalmol Vis Sci. 2013 Jan 2;54(1):9-18. doi: 10.1167/iovs.12-10241. PMID 23154459